CLINICAL TRIAL: NCT02958982
Title: A Phase I/IIa, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Safety, and Pharmacokinetics of Single and Multiple Ascending Dose of RP3128 in HV and Effect on LAR to Allergen Challenge in Mild Asthmatics
Brief Title: Safety, Tolerability and Pharmacokinetics of Oral Doses of RP3128 of Rhizen Pharmaceuticals
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Significant recruitment delay in POC part
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RP3128-1601
Record Dates: First submitted 2016-10-31; First posted 2016-11-08 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers; Asthma
Keywords: RP3128; Phase 1; Healthy volunteers
MeSH Terms: conditions — Asthma | interventions — RP3128

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RP3128 (Experimental): RP3128, A CRAC channel modulator
  Interventions: Drug: RP3128
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RP3128 — Participants will receive single oral dose of RP3128 in SAD, multiple dose in MAD AND POC
  Other Names: CRAC channel modulator
  Arms: RP3128
Drug: Placebo — Participants will receive single oral dose of RP3128 in SAD, multiple dose in MAD AND POC
  Arms: Placebo

SUMMARY:
RP3128 is a calcium release activated calcium (CRAC) channel modulator. The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of single and multiple ascending dose(s) of RP3128 in healthy volunteers and to evaluate the effect on late phase asthmatic response to allergen challenge in patients with mild asthma.

DETAILED DESCRIPTION:
The study consists of three parts; Part 1: single ascending dose (SAD), Part 2: multiple ascending dose (MAD) in healthy volunteers and Part 3: proof of concept (POC) study in mild asthmatics. There will be 5 cohorts in SAD and 3 cohorts in MAD, the doses used in the MAD will be based on emerging safety, tolerability and pharmacokinetics (PK) from Part 1 (SAD). POC is a randomized, placebo- controlled, double blind, two period cross-over, proof of concept study in male and female of non child bearing potential with history of mild asthma. the highest identified dose of RP3128 in Part 2 (MAD) will be considered for POC

ELIGIBILITY:
Inclusion Criteria:

* Male and non-childbearing female subjects (SAD/MAD) and male and non-childbearing female patients with mild asthma;
* Healthy subjects as determined by past medical history, vitals, physical examination and 12-lead ECG, clinical laboratory tests.
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive, weight ≥50 kg;
* Non-smokers or ex-smokers
* Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the subject; able to comply with protocol requirements and or study procedure;
* Negative screen for drugs of abuse and alcohol at screening and on admission.
* Male subjects should agree not to donate sperm for 3 months post dose; and
* Female partners (of child bearing potential) of male subjects should use 2 methods of highly effective contraception for 3 months post last

Additionally for POC

* Pre- bronchodilator Forced expiratory volume in 1 sec( FEV1) of > 70% (adjusted for age, sex and race)
* Steroid naïve subjects with history of mild asthma that satisfy the Global Initiative for Asthma (GINA) definition of asthma, but otherwise healthy.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant medical history.
* History of tuberculosis (TB) and/or a positive Tuberculin Skin Test and/or QuantiFeron- TB®-Gold test.
* Use of any immunotherapy within 3 months prior to screening.
* History of serious adverse reaction, severe hypersensitivity or allergy to any drug/drug substance (except house dust mite, pollen allergens or cat dander allergy in asthmatics) or in any other circumstance (e.g. anaphylaxis);
* Abnormal liver function
* Positive screen on hepatitis-B surface antigen (HBsAg), antibodies to the hepatitis C (HCV) or antibodies to the human immunodeficiency virus (HIV) 1,2;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inflamax Research Inc., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barde PJ, Viswanadha S, Veeraraghavan S, Vakkalanka SV, Nair A. A first-in-human study to evaluate the safety, tolerability and pharmacokinetics of RP3128, an oral calcium release-activated calcium (CRAC) channel modulator in healthy volunteers. J Clin Pharm Ther. 2021 Jun;46(3):677-687. doi: 10.1111/jcpt.13322. Epub 2020 Dec 11. PMID 33314326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 03 Nov 2016 to 05 Apr 2017 for Single Ascending Dose (SAD) study and patients were recruited between 12 May 2017 to 26 Aug 2017 for Multiple Ascending Dose (MAD) study
Pre-assignment Details: There are only two groups: RP3128 and Placebo. Since this is a dose escalation study, the healthy volunteers enrolled in each cohorts are combined together and presented as study drug (RP3128) and Placebo (SAD and MAD). The proof of concept study was terminated prematurely after enrolling only one patient. Therefore, no analysis was performed.
Groups:
- Pooled Placebo (SAD): Placebo
  Placebo: Participants will receive single oral dose of RP3128 in SAD,
- RP3128_25 mg_SAD: Participants will receive single oral dose of 25 mg of RP3128 once a day in SAD
- RP3128_50 mg_SAD: Participants will receive single oral dose of 50 mg of RP3128 once a day in SAD
- RP3128_100 mg_SAD: Participants will receive single oral dose of 100 mg of RP3128 once a day in SAD
- RP3128_200 mg_SAD: Participants will receive single oral dose of 200 mg of RP3128 once a day in SAD
- RP3128_400 mg_SAD: Participants will receive single oral dose of 400 mg of RP3128 once a day in SAD
- Pooled Placebo (MAD): Placebo
  Placebo: Participants will receive single oral dose of RP3128 in MAD,
- RP3128_25 mg_MAD: Participants will receive multiple oral dose of 25 mg of RP3128 for a week in MAD,
- RP3128_100 mg_MAD: Participants will receive multiple oral dose of 100 mg of RP3128 for a week in MAD,
- RP3128_400 mg_MAD: Participants will receive multiple oral dose of 400 mg of RP3128 for a week in MAD,
- Proof of Concept: RP3128/Placebo
Period: Cohort 1: 25 mg in SAD Study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Started | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: 50 mg in SAD Study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Started | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3: 100 mg in SAD Study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Started | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 4: 200 mg in SAD Study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Started | 2 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 5: 400 mg in SAD Study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Started | 2 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1 : 25 mg in MAD Study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: 100 mg in MAD Study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3: 400 mg in MAD Study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Proof of Concept Study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Since this is a dose escalation study, the healthy volunteers enrolled in each cohorts are combined together and presented as study drug (RP3128) and Placebo for, the baseline characteristics and outcomes in both SAD and MAD. Since the POC study terminated, one patient who recruited in POC was not considered for baseline measures
Groups:
- Pooled Placebo (SAD): Placebo: Participants will receive single oral dose of Placebo in SAD
- RP3128_25 mg_SAD: RP3128: Participants will receive single oral dose of 25 mg of RP3128 in SAD
- RP3128_50 mg_SAD: RP3128: Participants will receive single oral dose of 50 mg of RP3128 in SAD
- RP3128_100 mg_SAD: RP3128: Participants will receive single oral dose of 100 mg of RP3128 in SAD
- RP3128_200 mg_SAD: RP3128: Participants will receive single oral dose of 200 mg of RP3128 in SAD
- RP3128_400 mg_SAD: RP3128: Participants will receive single oral dose of 400 mg of RP3128 in SAD
- Pooled Placebo: Placebo: Participants will receive multiple oral doses of placebo in MAD
- RP3128_25 mg_MAD: RP3128: Participants will receive multiple oral dose of 25 mg of RP3128 in MAD
- RP3128_100 mg_MAD: RP3128: Participants will receive multiple oral dose of 100 mg of RP3128 in MAD
- RP3128_400 mg_MAD: RP3128: Participants will receive multiple oral dose of 400 mg of RP3128 in MAD
- Proof of Concept: Patient received at least one dose of RP3128/placebo
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept | Total
Number analyzed (Participants) | 9 | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 8 | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.4 (8.26) | 36.3 (4.93) | 36.3 (9.07) | 31.5 (6.61) | 38.2 (8.30) | 34.7 (9.42) | 36.7 (4.59) | 29.5 (6.92) | 33.2 (3.43) | 36.5 (5.39) | 32.0 (0) | 33.6 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 9 | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 0 | 1 | 0 | 1 | 3 | 3 | 2 | 0 | 16
  Not Hispanic or Latino | 7 | 0 | 3 | 4 | 5 | 6 | 5 | 3 | 3 | 4 | 1 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 2 | 4 | 2 | 1 | 2 | 1 | 0 | 15
  White | 6 | 2 | 2 | 3 | 3 | 2 | 3 | 5 | 3 | 4 | 0 | 33
  More than one race | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment
Time Frame: Baseline through 2 weeks
Population: There are only two groups: RP3128 and Placebo. Since this is a dose escalation study, the healthy volunteers enrolled in each cohorts are combined together and presented as study drug (RP3128) and Placebo for, the baseline characteristics and outcomes in both SAD and MAD.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo (SAD): Placebo: Participants will receive single oral dose of RP3128 in SAD,
- Pooled Placebo (MAD): Placebo: Participants will receive single oral dose of RP3128 in MAD,
- RP3128_25 mg_MAD: RP3128 (MAD): Participants will receive multiple oral dose of 25 mg of RP3128 in MAD,
- RP3128_100 mg_MAD: RP3128 (MAD): Participants will receive multiple oral dose of 100 mg of RP3128 in MAD study
- RP3128_400 mg_MAD: RP3128 (MAD): Participants will receive multiple oral dose of 400 mg of RP3128 in MAD study
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Number analyzed (Participants) | 9 | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Participants | 4 | 1 | 2 | 4 | 2 | 4 | 3 | 1 | 0 | 2 | 0

2. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: Cmax after administration of RP3128/ placebo in part 1 and part 2
Time Frame: Pre-dose through 48 hours post dose
Measure: Mean (Standard Deviation); unit: micrograms/mL
Groups:
- RP3128_25 mg_SAD: RP3128: Participants will receive single oral dose of 25 mg RP3128 in SAD (Day1)
- RP3128_50 mg_SAD: RP3128: Participants will receive single oral dose of 50 mg RP3128 in SAD (Day1)
- RP3128_100 mg_SAD: RP3128: Participants will receive single oral dose of 100 mg RP3128 in SAD (Day1)
- RP3128_200 mg_SAD: RP3128: Participants will receive single oral dose of 200 mg RP3128 in SAD (Day1)
- RP3128_400 mg_SAD: RP3128: Participants will receive single oral dose of 400 mg RP3128 in SAD (Day1)
- RP3128_25 mg_MAD: RP3128 (MAD): Participants will receive multiple oral dose of 25 mg of RP3128 in MAD (Day 7),
- RP3128_100 mg_MAD: RP3128 (MAD): Participants will receive multiple oral dose of 100 mg of RP3128 in MAD (Day 7),
- RP3128_400 mg_MAD: RP3128 (MAD): Participants will receive multiple oral dose of 400 mg of RP3128 in MAD (Day 7),
- Proof of Concept: Participants will RP3128/Placebo
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Number analyzed (Participants) | 9 | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 1
micrograms/mL | 0 (0) | 0.171 (0.041) | 0.305 (0.075) | 0.561 (0.12) | 0.64 (0.29) | 0.915 (0.41) | 0 (0) | 0.533 (0.10) | 2.034 (1.11) | 3.95 (2.16) | 0 (0)

3. Secondary Outcome: Measurement of Cytokines
Description: Levels of cytokines following LPS (lipopolysaccharide) or CD3/CD28 stimulation.
Time Frame: Predose and Day 7 in Part 2
Reporting Status: Not Posted

4. Secondary Outcome: Fractional Exhaled Nitric Oxide (FeNo)
Description: Change in FeNo after administration of RP3128/ placebo in part 3
Time Frame: Prechallenge to 3, 8 and 24 hours post challenge in Part 3
Reporting Status: Not Posted

5. Secondary Outcome: Area Under Effective Concentration (AUEC)
Description: AUEC0-3h, AUEC3-8h after administration of RP3128/ placebo in part 3
Time Frame: 0 to 3 hours and 3 to 8 hours post allergen challenge in Part 3
Reporting Status: Not Posted

6. Secondary Outcome: Cell Count
Description: Absolute and % counts of sputum eosinophils and neutrophils
Time Frame: 8 and 24 hours post allergen challenge in Part 3
Reporting Status: Not Posted

7. Secondary Outcome: Area Under the Plasma-Concentration
Description: AUC0-t after administration of RP3128/ placebo in part 1 and part 2
Time Frame: Pre-dose through 48 hours post dose
Measure: Mean (Standard Deviation); unit: micrograms*hours/mL
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
Number analyzed (Participants) | 9 | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 1
micrograms*hours/mL | 0 (0) | 8.821 (0.47) | 10.766 (3.884) | 30.340 (9.968) | 37.011 (14.56) | 94.227 (39.29) | 0 (0) | 7.934 (1.23) | 31.034 (19.71) | 61.821 (39.023) | 0 (0)

ADVERSE EVENTS:
Time Frame: 15 Days
Description: There are only two groups: RP3128 and Placebo. Since this is a dose escalation study, the healthy volunteers enrolled in each cohorts are combined together and presented as study drug (RP3128) and Placebo for, the baseline characteristics and outcomes in both SAD and MAD
Groups:
- RP3128_25 mg_SAD: RP3128: Participants will receive single oral dose 25 mg of RP3128 in SAD
- RP3128_50 mg_SAD: RP3128: Participants will receive single oral dose 50 mg of RP3128 in SAD
- RP3128_100 mg_SAD: RP3128: Participants will receive single oral dose 100 mg of RP3128 in SAD
- RP3128_200 mg_SAD: RP3128: Participants will receive single oral dose 200 mg of RP3128 in SAD
- RP3128_400 mg_SAD: RP3128: Participants will receive single oral dose 400 mg of RP3128 in SAD
- RP3128_25 mg_MAD: RP3128 (MAD): Participants will receive multiple oral dose 25 mg of RP3128 for one week in MAD,
- RP3128_100 mg_MAD: RP3128 (MAD): Participants will receive multiple oral dose 100 mg of RP3128 for one week in MAD,
- RP3128_400 mg_MAD: RP3128 (MAD): Participants will receive multiple oral dose 400 mg of RP3128 for one week in MAD,
- Proof of Concept: Participants will receive RP3128/Placebo
Arm/Group | Pooled Placebo (SAD) | RP3128_25 mg_SAD | RP3128_50 mg_SAD | RP3128_100 mg_SAD | RP3128_200 mg_SAD | RP3128_400 mg_SAD | Pooled Placebo (MAD) | RP3128_25 mg_MAD | RP3128_100 mg_MAD | RP3128_400 mg_MAD | Proof of Concept
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/1
Other Adverse Events (participants affected / at risk) | 4/9 | 1/3 | 2/4 | 4/4 | 2/6 | 4/6 | 3/6 | 1/6 | 0/6 | 2/6 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (SAD) (N=9) | RP3128_25 mg_SAD (N=3) | RP3128_50 mg_SAD (N=4) | RP3128_100 mg_SAD (N=4) | RP3128_200 mg_SAD (N=6) | RP3128_400 mg_SAD (N=6) | Pooled Placebo (MAD) (N=6) | RP3128_25 mg_MAD (N=6) | RP3128_100 mg_MAD (N=6) | RP3128_400 mg_MAD (N=6) | Proof of Concept (N=1)
General disorders (General disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Disorders (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations (Investigations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders (Nervous system disorders) | 1 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
There is no limitations and Caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT02958982/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02958982/SAP_001.pdf